CLINICAL TRIAL: NCT03018158
Title: MR Images Variation With or Without Denture Wear. Motion Artifacts Related With Tongue Movements
Brief Title: MR Images Variation With or Without Denture Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nihon University (Other)
Responsible Party: Principal Investigator, Yasuhiko Kawai, Professor Dr.Yasuhiko kawai, Nihon University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EC 15-019
Record Dates: First submitted 2016-12-28; First posted 2017-01-11 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Magnetic Resonance Imaging
MeSH Terms: interventions — Dental Restoration Wear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- dentulous (No Intervention): MR Imaging was collected with condition at the tongue at rest position.
- edentulous without denture wear. (No Intervention): MR Imaging was collected without denture wear.
- edentulous with denture wear. (Experimental): MR Imaging was collected with denture wear.
  Interventions: Device: denture wear.

INTERVENTIONS:
Device: denture wear. — MR Imaging was collected with or without denture wear.
  Arms: edentulous with denture wear.

SUMMARY:
The objective of this study was to compare level of artifact while tongue at rest and in motion of dentulous subjects.

DETAILED DESCRIPTION:
The magnetic resonance imaging (MRI) is useful to diagnose soft tissue morphology, especially to detect cancer and disk displacement with temporomandibular disorders. The prevalence of tongue cancer may increase with ageing population. A clear MR image is indispensable for clinical diagnosis. However, tongue motion associated with the habitual or swallowing tongue movement may cause artifacts on MRI. This occurrence of motion artifact is speculated to be prominent with the patients without the occlusal support. The objective of this pilot study was to compare level of artifact while tongue at rest and in motion of dentulous subjects.

ELIGIBILITY:
Inclusion Criteria:

* dentulous
* edentulous classified Eichner' s classfication

Exclusion Criteria:

* involuntary motion occurs during imaging
* absolutely contraindicated or as a rule contraindicated of MRI examination
* subjects have ferromagnetic metals in the oral cavity
* subjects can not swallow naturally

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Luminance standard deviation value on MR image | MR Imaging was collected with each condition.Through study completion, an average of 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiko Kawai, DDS MSc PhD, Study Chair — Nihon University
Locations (1):
- Nihon University Hospital, Matsudo, Chiba, Japan

IPD SHARING:
Plan to Share IPD: No